CLINICAL TRIAL: NCT03998280
Title: The Effect of Cervical Muscle Fatigue on Neck Proprioception and Postural Stability
Brief Title: The Effect Of Cervical Muscle Fatigue in Neck Proprioception and Postural Stability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alaa Yousri Mahmoud Atia (Other Government)
Responsible Party: Sponsor-Investigator, Alaa Yousri Mahmoud Atia, physiotherapest, Ministry of Health and Population, Egypt
Organization: Ministry of Health and Population, Egypt (Other Government)
Other Study IDs: P. T. REC/012/002299
Record Dates: First submitted 2019-06-14; First posted 2019-06-26 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Muscle Fatigue
Keywords: fatigue ,deep neck flexor
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Assessment — Neck proprioception and postural stability

SUMMARY:
PURPOSE:

To investigate the effect of cervical muscle Fatigue on neck proprioception and postural stability during cervical flexion.

BACKGROUND:

Postural stability is the ability to maintain the body in equilibrium either at rest or in a steady state of motion . Muscle fatigue is the diminished response of muscle to repeated stimulus. Cervical proprioceptive inputs provide important somatosensory information influencing postural stability. Hence, the investigators performed this study to evaluate the effect of experimentally induced fatigue on general cervical musculature on postural stability .

HYPOTHESES:

This study will hypnotize that:

1. Cervical flexor muscle fatigue will have a significant effect on neck proprioception
2. Cervical muscle fatigue will have a significant effect on posture stability

RESEARCH QUESTION:

Will fatigue of cervical flexors have an effect on neck proprioception and postural stability?

DETAILED DESCRIPTION:
the research methodology that will be used

Induction of fatigue using isometric neck flexor muscle endurance test (NET):

An isometric neck muscle endurance test (NME test) will be performed for the deep neck flexors (Rectus Capitus Anterior, Rectus Capitus Lateralis, Longus Capitus, Longus Colli) until exhaustion in all participants occurs. With the subject in hook lying position through CHIN RETRACTION AND HEAD ELEVATED FROM THE COUCH.

All the assessment measurements will be done before and just immediately after performing the cervical muscle fatigue then after 15 minutes of fatigue induction(fatigue recovery) A. Measurement of neck proprioception using cervical joint position error test via OVERHEAD LASER POINTER

B. Measurement of postural stability using :

1. Biodex balance system(limit of stability) to measure postural stability
2. Multi-Directional Reach Test

ELIGIBILITY:
Inclusion Criteria:

* having cervical range of motion 80 to 90 of flextion, 70 degree of extension, 20 to 45 degrees if lateral flextion, and 80 to 90 rotation to both sides.
* having normaluscle test strength for cervical neck flexors according to group manual muscle test
* body mass index ranging from 18.5 to 24.9 kg/m2

Exclusion Criteria:

* any history of pathological truma to the cervical,thoracic or lumbar spine, upper extremity or rib cage.
* surgical condition of the spine
* having any orthopedic, musculoskeletal or neurological disorders around cervical region.
* any vestibular impairment (e.g.vertigo)
* spinal postural deformities as hyper kyphosis &scoliosis

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Residents from certain town
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-03-31 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-20 (Estimated)

PRIMARY OUTCOMES:
Induction of fatigue using isometric neck flexor muscle endurance test (NET): | six months
  a. An isometric neck muscle endurance test (NME test) will be performed for the deep neck flexors (Rectus Capitus Anterior, Rectus Capitus Lateralis, Longus Capitus, Longus Colli) until exhaustion in all participants occurs. with the subject in hook lying position through CHIN RETRACTION AND HEAD ELEVATED FROM THE COUCH.

SECONDARY OUTCOMES:
Measurement of neck proprioception using cervical joint position error test via OVERHEAD LASER POINTER | six months
  : A laser pointer will be fixed to a headband or strap. Target paper will be typically 40 cm in diameter that contains concentric circles in 1 cm increments, divided into 4 quadrants intersecting at the zero.

OTHER OUTCOMES:
Multi-Directional Reach Test | six months
  Multi-Directional Reach (MDRT) is an inexpensive screening tool to determine the limits of stability of individuals in 4 directions. It measure how far an individual can voluntarily reach, thereby shifting the COG to the limits of the BOS with the feet stationary. The MDRT is a valid and reliable clinical measure for limits of stability. The test can be used to assess human postural stability in different four direction as follow (Roberta 2001)
Biodex Balance System for The postural stability test | six months
  The postural stability test emphasized on subject's ability to maintain center of balance. The subject's score on this test will assess the deviations from center, thus a lower score is more desirable than a higher score. Platform stability could be varied during this test by selecting (more options) from the Postural Stability Testing screen. It was proved that trial time, number of trials, starting and ending platform stability, rest count-downs or bilateral test could be set (Tropp and Odenrick., 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided